CLINICAL TRIAL: NCT03716999
Title: Starlight Therapy as a Non-Pharmacological Nursing Intervention in Palliative Care
Brief Title: Starlight Therapy in Palliative Care
Status: Not yet recruiting | Type: Observational
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Other Study IDs: Starlight Trial
Record Dates: First submitted 2018-10-18; First posted 2018-10-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-02

CONDITIONS: Symptom Management
Keywords: palliative; starlight; end-of-life symptoms; non-pharmacological

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Palliative Care Patients: Palliative care Patients meeting criteria will receive Starlight Therapy
  Interventions: Other: Starlight Therapy

INTERVENTIONS:
Other: Starlight Therapy — Starlight Projector will be placed in patients' rooms and project starlight on the ceilings and walls in an effort to reduce unpleasant symptoms

SUMMARY:
Starlight Therapy™ has been shown to help alleviate end-of-life symptoms in Palliative Care patients and reduce the need for PRN or "as needed" medications. This study will investigate the efficacy of this intervention on the symptom of anxiety using a mixed-method analysis.

The primary investigator hypothesizes that any anti-anxiolytic effects could be caused by the Intrinsically Photosensitive Retinal Ganglion Cell neural pathway to the amygdala.

DETAILED DESCRIPTION:
Starlight Therapy has been shown (see citation) to help alleviate end-of-life symptoms in Palliative Care patients and reduce the need for PRN or "as needed" medications. This study will investigate the efficacy of this intervention using a mixed-method analysis.

Starlight Therapy will be offered to patients with unpleasant end-of-life symptoms such as dyspnea, agitation, anxiety, restlessness and insomnia. The effect the Starlight Therapy has in helping alleviate these symptoms will be measured using the ESAS (Edmonton Symptom Assessment System) questionnaire at baseline and following a predetermined period of time of Starlight Therapy.

10 Starlight Projectors have been purchased for the unit where the study will take place: the Inpatient Palliative Care Unit 7A, Victoria General Hospital, Centennial Building. The funding was acquired by a Comfort & Care Grant from the QEII Foundation.

The results will be compiled and analyzed in a research paper "Concerning the Efficacy and Underlying Mechanism of Starlight Therapy as a Non-Pharmacological Nursing Intervention for Palliative Care Patients".

ELIGIBILITY:
Inclusion Criteria:

1. ESAS indicates at least one of the following symptoms:

* Insomnia
* Anxiety
* Restlessness
* Dyspnea
* Pain

Exclusion Criteria:

1. Clinical Diagnosis of blindness
2. ESAS does not include any of the flowing symptoms:

   * Insomnia
   * Anxiety
   * Restlessness
   * Dyspnea
   * Pain

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients in an inpatient palliative care Setting who meet the specified criteria for inclusion in the study
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-12-15 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Using Starlight Therapy to measure Change in Unpleasant Symptoms in Palliative Care Patients as measured using the ESAS (Edmonton Symptom Assessment System) Scale. On a scale of 0-10, with 0 = no symptom and 10= symptom is worst outcome possible. | 2 hours of Starlight Therapy
  Edmonton Assessment scale questionnaire will be completed before Starlight Therapy and after 2 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Victoria General Hospital, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Evaluation of a Low-Light Intervention-Starlight Therapy-for Agitation, Anxiety, Restlessness, Sleep Disturbances, Dyspnea, and Pain at End of Life. (2017). Journal of Hospice & Palliative Nursing, 19(3), 221-222. doi:10.1097/njh.0000000000000343
- See also: Quantitative study on Starlight Therapy — https://journals.lww.com/jhpn/Citation/2017/06000/Evaluation_of_a_Low_Light_Intervention_Starlight.7.aspx